CLINICAL TRIAL: NCT03208153
Title: Randomized Comparison Between the Invasive and Conservative Strategies in Elderly Frail Patients With Non-ST Elevation Myocardial Infarction: The MOSCA-FRAIL Clinical Trial
Brief Title: the Invasive and Conservative Strategies in Elderly Frail Patients With Non-STEMI
Acronym: MOSCA-FRAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Spanish Society of Cardiology (Other); Instituto de Investigacion Sanitaria INCLIVA (Other)
Responsible Party: Principal Investigator, Juan Sanchis, Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOSCA-II
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Non-ST Elevation Myocardial Infarction; Frail Elderly Syndrome
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Invasive (Experimental): In-hospital routine coronary angiogram and revascularization if anatomically feasible
  Interventions: Procedure: Invasive
- Conservative (Active Comparator): In-hospital coronary angiogram only if poor clinical course
  Interventions: Procedure: Conservative

INTERVENTIONS:
Procedure: Invasive — Coronary angiogram and revascularization if anatomically feasible
  Arms: Invasive
Procedure: Conservative — Conservative
  Arms: Conservative

SUMMARY:
The role of a routine invasive strategy in frail patients with non-ST-segment elevation acute myocardial infarction is currently uncertain. We hypothesize that a routine invasive strategy will improve outcomes. The aim of the trial is to evaluate the efficacy and safety of a routine invasive strategy in increasing the number of days alive at home during the first year and improving cardiovascular outcomes.

DETAILED DESCRIPTION:
There is a lack of evidence for the best management of frail patients with non-ST-elevation myoardial infaarction (NSTEMI). Clinical practice guidelines recommend a routine invasive strategy in NSTEMI in the majority of patients (Roffi Eur Heart 2016). Nevertheless, invasive management is underused in frail and patients with comorbidity (Ekerstad Circulation 2011, Sanchis Mayo Clin Proceed 2011, Graham Can J Cardiol 2013,). Furthermore, frail patients undergoing coronary angiography have lower revascularisation rates than non frail counterparts (Ekerstad Circulation 2011, Graham Can J Cardiol 2013). This may be, in part, a reflection of the more complex coronary artery disease, more frequently presenting left main, three vessel disease or proximal coronary artery disease, which may not be amenable to PCI (Singh Circ Cardiovasc Qualit Outco 2011). However, it is also possible that lower rates reflect an aversion to a perceived risk of the intervention in the frail, whereby those with potential to gain benefit may have been deemed not appropriate for coronary intervention. After PCI or cardiac surgery, frailty and comorbidity are associated with adverse long-term outcomes (Singh CircQualitOutco 2011, SundermanEur J Cardio-thoracic Surgery 2011). Comorbid patients, however, could benefit the most from in-hospital revascularization in NSTEMI (Bauer et al Eur Heart J 2007, Palau Clin Cardiol 2012).

A few studies addressed the role of invasive strategy in elderly patients. A routine invasive strategy was not statistically superior to a selective invasive strategy in elderly patients with NSTEMI (Savonito JACC CIV 2012) but the study was underpowered due to the small sample size. The After Eighty randomized trial was a proper-sized study which included patients >80 years with NSTEMI and demonstrated the benefit of the invasive strategy in reducing the composite endpoint of death or cardiovascular events at 1.5 years (Tegn Lancet 2016). It is worth noting that no patient underwent cardiac catheterization under any circumstance in the conservative arm of that study. Furthermore, only 23% of the potential candidates for inclusion were finally randomized, suggesting a bias towards lower risk patients, a very restrictive approach. Recently, the MOSCA randomized trial evaluated the efficacy of an invasive strategy in elderly patients with NSTEMI and comorbidities (Sanchis Eur J Intern Med 2016). Although this was a small trial, the invasive strategy reduced the probability of death or ischemic events at 3 months. This benefit, nonetheless, vanished at 2.5-years follow-up. No clinical trials specifically designed to investigate the management of frail patients in NSTEMI have been conducted so far. In fact, frail patients have usually been excluded from randomized clinical trials. The TRILOGY-ACS trial, for instance, included a remarkably low rate (4.7%) of frail patients (White, Eur Heart J ACC 2016).

On the other hand, while most of the studies mainly focus on death, myocardial infarction, stroke, need for revascularisation or rehospitalisation, patients are also willing to recover an independent life and return to their usual place for living. The presence of geriatric syndromes (including frailty, cognitive impairment, severe dependence and depression) is not only associated with worse clinical outcomes but with a greater risk of functional decline and need for new social help, that is an increased level of dependence. This has an important impact on the patient quality of life and psychological wellbeing but also frequently becomes a heavy social and economic burden for patients and families. Therefore, one of the real challenges in the management of ACS in very old patients is the prevention of dependence. In this sense, the use of new outcomes especially addressed to measure level of independence and quality of life is especially important (Montilla I, Heart Lung Circ 2016).

The role of a routine invasive strategy in frail patients is currently uncertain. We hypothesize that a routine invasive strategy in frail patients with NSTEMI will improve outcomes. The aim of the trial is to evaluate the efficacy and safety of a routine invasive strategy in increasing the number of days alive at home during the first year and improving cardiovascular outcomes. A prespecified subgroup analysis will be conducted according to comorbidities and Charlson index

ELIGIBILITY:
Inclusion Criteria:

* Non-ST-elevation acute myocardial infarction
* Age ≥70 years
* Frailty criteria defined by =>4 points in the Clinical Frailty Scale (Rockwood K CMAJ 2005).

Exclusion Criteria:

* Prior known non-revascularizable coronary artery disease
* Significant concomitant non-ischemic heart disease (i.e. severe heart valve disease, hypertrophic cardiomyopathy…)
* Unable to understand/sign informed consent
* Life expectancy <12 months

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 167 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
number of days alive out of the hospital | 1 year
  number of days alive out of the hospital
major adverse cardiac events | 1 year
  cardiovascular death or myocardial infarction or revascularization

SECONDARY OUTCOMES:
all-cause death | 1 and 3 years
cardiovascular death | 1 and 3 years
myocardial infarction | 1 and 3 years
rehospitalization for cardiac and extra-cardiac causes | 1 and 3 years
bleeding episodes | 1 and 3 years
stroke | 1 and 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic Hospital, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Result] Savonitto S, Cavallini C, Petronio AS, Murena E, Antonicelli R, Sacco A, Steffenino G, Bonechi F, Mossuti E, Manari A, Tolaro S, Toso A, Daniotti A, Piscione F, Morici N, Cesana BM, Jori MC, De Servi S; Italian Elderly ACS Trial Investigators. Early aggressive versus initially conservative treatment in elderly patients with non-ST-segment elevation acute coronary syndrome: a randomized controlled trial. JACC Cardiovasc Interv. 2012 Sep;5(9):906-16. doi: 10.1016/j.jcin.2012.06.008. PMID 22995877
- [Result] Tegn N, Abdelnoor M, Aaberge L, Endresen K, Smith P, Aakhus S, Gjertsen E, Dahl-Hofseth O, Ranhoff AH, Gullestad L, Bendz B; After Eighty study investigators. Invasive versus conservative strategy in patients aged 80 years or older with non-ST-elevation myocardial infarction or unstable angina pectoris (After Eighty study): an open-label randomised controlled trial. Lancet. 2016 Mar 12;387(10023):1057-1065. doi: 10.1016/S0140-6736(15)01166-6. Epub 2016 Jan 13. PMID 26794722
- [Result] Sanchis J, Nunez E, Barrabes JA, Marin F, Consuegra-Sanchez L, Ventura S, Valero E, Roque M, Bayes-Genis A, Del Blanco BG, Degano I, Nunez J. Randomized comparison between the invasive and conservative strategies in comorbid elderly patients with non-ST elevation myocardial infarction. Eur J Intern Med. 2016 Nov;35:89-94. doi: 10.1016/j.ejim.2016.07.003. Epub 2016 Aug 8. PMID 27423981
- [Result] Nunez J, Ruiz V, Bonanad C, Minana G, Garcia-Blas S, Valero E, Nunez E, Sanchis J. Percutaneous coronary intervention and recurrent hospitalizations in elderly patients with non ST-segment acute coronary syndrome: The role of frailty. Int J Cardiol. 2017 Feb 1;228:456-458. doi: 10.1016/j.ijcard.2016.11.151. Epub 2016 Nov 10. No abstract available. PMID 27870976
- [Result] Sanchis J, Ruiz V, Bonanad C, Valero E, Ruescas-Nicolau MA, Ezzatvar Y, Sastre C, Garcia-Blas S, Mollar A, Bertomeu-Gonzalez V, Minana G, Nunez J. Prognostic Value of Geriatric Conditions Beyond Age After Acute Coronary Syndrome. Mayo Clin Proc. 2017 Jun;92(6):934-939. doi: 10.1016/j.mayocp.2017.01.018. Epub 2017 Apr 25. PMID 28389067
- [Derived] Sanchis J, Bueno H, Marti Sanchez D, Martinez-Selles M, Diez Villanueva P, Barrabes JA, Marin F, Villa A, Sanmartin Fernandez M, Llibre C, Sionis A, Elizaga J, Alfonso F, Nunez E, Nunez J, Kunadian V, Ariza-Sole A. Effects of routine invasive management on reinfarction risk in older adults with frailty and non-ST-segment elevation myocardial infarction: a subanalysis of a randomised clinical trial. Heart. 2025 Jul 28;111(16):786-792. doi: 10.1136/heartjnl-2024-325254. PMID 39922692
- [Derived] Sanchis J, Bueno H, Garcia-Blas S, Alegre O, Marti D, Martinez-Selles M, Dominguez-Perez L, Diez-Villanueva P, Barrabes JA, Marin F, Villa A, Sanmartin M, Llibre C, Sionis A, Carol A, Fernandez-Cisnal A, Calvo E, Morales MJ, Elizaga J, Gomez I, Alfonso F, Garcia Del Blanco B, Formiga F, Nunez E, Nunez J, Ariza-Sole A. Invasive Treatment Strategy in Adults With Frailty and Non-ST-Segment Elevation Myocardial Infarction: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Mar 4;7(3):e240809. doi: 10.1001/jamanetworkopen.2024.0809. PMID 38446482
- [Derived] Sanchis J, Bueno H, Minana G, Guerrero C, Marti D, Martinez-Selles M, Dominguez-Perez L, Diez-Villanueva P, Barrabes JA, Marin F, Villa A, Sanmartin M, Llibre C, Sionis A, Carol A, Garcia-Blas S, Calvo E, Morales Gallardo MJ, Elizaga J, Gomez-Blazquez I, Alfonso F, Garcia Del Blanco B, Nunez J, Formiga F, Ariza-Sole A. Effect of Routine Invasive vs Conservative Strategy in Older Adults With Frailty and Non-ST-Segment Elevation Acute Myocardial Infarction: A Randomized Clinical Trial. JAMA Intern Med. 2023 May 1;183(5):407-415. doi: 10.1001/jamainternmed.2023.0047. PMID 36877502
- [Derived] Sanchis J, Ariza-Sole A, Abu-Assi E, Alegre O, Alfonso F, Barrabes JA, Baz JA, Carol A, Diez Villanueva P, Garcia Del Blanco B, Elizaga J, Fernandez E, Garcia Del Egido A, Garcia Picard J, Gomez Blazquez I, Gomez Hospital JA, Hernandez-Antolin R, Llibre C, Marin F, Marti Sanchez D, Martin R, Martinez Selles M, Minana G, Morales Gallardo MJ, Nunez J, Perez de Prado A, Pinar E, Sanmartin M, Sionis A, Villa A, Marrugat J, Bueno H. Invasive Versus Conservative Strategy in Frail Patients With NSTEMI: The MOSCA-FRAIL Clinical Trial Study Design. Rev Esp Cardiol (Engl Ed). 2019 Feb;72(2):154-159. doi: 10.1016/j.rec.2018.02.007. Epub 2018 Mar 7. English, Spanish. PMID 29525724